CLINICAL TRIAL: NCT03791684
Title: Accelerated Versus Standard Corneal Cross Linking in the Treatment of Ectasia Post Refractive Surgery and Penetrating Keratoplasty: A Long Term Randomized Trial.
Brief Title: Accelerated Versus Standard CXL in the Treatment of Ectasia Post Refractive Surgery and Penetrating Keratoplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hany Khairy, Consultant Ophthalmology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ophth001/2016
Record Dates: First submitted 2018-12-24; First posted 2019-01-03 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Refractive Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated Cross Linking (Active Comparator): Ultraviolet A radiation of 365 nm wavelength (CCL-365 vario, Peschke Meditrade GmbH, Switzerland), and an irradiance of 18mW/cm2 (spot size 7mm), at a distance of 45 mm from the cornea, was applied for a period of 5 min, delivering a dose of 5.4 J/cm2.
  Interventions: Device: Cross linking
- Standard Cross linking (Active Comparator): Ultraviolet A radiation of 365 nm wavelength (CCL-365 vario, Peschke Meditrade GmbH, Switzerland), and an irradiance of 3mW/cm2 (spot size 7mm), at a distance of 45 mm from the cornea, was applied for a period of 30 min, delivering a dose of 5.4 J/cm2.
  Interventions: Device: Cross linking

INTERVENTIONS:
Device: Cross linking — Cross linking strategy either standard or accelerated

SUMMARY:
WHAT WAS KNOWN

*Standard CXL is the common procedure for treating progressive corneal ectasia. Modifications of the standard protocol were introduces to reduce its complications especially long exposure to ultraviolet rays. The Accelerated protocol, while believed to overcome this issue with comparable outcomes, has not been studied fully in patients with ectasia following corneal refractive surgery and penetrating keratoplasty.

WHAT THIS PAPER ADDS Accelerated CXL is as safe and effective as the Standard CXL in halting the progression of ectasia post refractive surgery and penetrating keratoplasty with the benefit of: reduced ultraviolet exposure, reduced operation time, and reduced patient discomfort.

DETAILED DESCRIPTION:
Purpose:

The aim of this study is to compare the clinical outcomes of the Standard CXL and the AC CXL in patients with progressive corneal ectasia post refractive surgery and penetrating keratoplasty.

Setting:

Menoufia University Hospital, Egypt

Design:

Prospective, randomised comparison.

Methods:

Patients scheduled to receive either Standard CXL (3mW/cm2 for a period of 30 min) or Accelerated CXL (18mW/cm2 for a period of 5 min).The main outcomes for comparison were the change in; Maximum-K reading (K-max), manifest refractive spherical equivalent (SE), central corneal thickness (CCT), and the best corrected distance visual acuity (CDVA).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were:
* adults aged above 18 years.
* They have been diagnosed clinically with progressive corneal ectasia following refractive surgery procedure (LASIK, PRK, ReLex smile), or penetrating keratoplasty
* CCT above 400µ.

Exclusion Criteria:

* The exclusion criteria involved:
* history of herpetic ocular diseases (including herpes simplex virus and varicella zoster virus) in the study eye
* active or recurrent ocular disease in either eye (e.g., uveitis, chronic moderate to severe blepharitis or severe dry eye) or sight-threatening diseases (e.g., previous retinal or optic nerve diseases) that would interfere with the interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
K-max changes | 12 post treatment
  The main outcomes for comparison were the change in; Maximum-K reading (K-max), Patients were followed up clinically on the first day, first week, one month, 6 months and 12 months postoperatively

SECONDARY OUTCOMES:
manifest refractive spherical equivalent (SE) in Diopter power | 12 months postoperatively
  The secondary outcomes for comparison were the change in, manifest refractive spherical equivalent (SE).
  Patients were followed up clinically on the first day, first week, one month, 6 months and 12 months postoperatively

IPD SHARING:
Plan to Share IPD: Yes
The data used to support the findings of this study are restricted by the Ophthalmic Ethics Committee at Menoufia University Hospital, in order to protect patient privacy. Data are available from Mr Hany Khairy (khairyhany@hotmail.com), for researchers who meet the criteria for access to confidential data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data used to support the findings of this study are restricted by the Ophthalmic Ethics Committee at Menoufia University Hospital, in order to protect patient privacy. Data are available from Mr Hany Khairy (khairyhany@hotmail.com), for researchers who meet the criteria for access to confidential data after study publcation
Access Criteria: Data are available for researchers who meet the criteria for access to confidential data as specified by the Ophthalmic Committee of Menoufia University Hospital